CLINICAL TRIAL: NCT01854710
Title: Thorough QT/QTc Study of 2 Doses of ADASUVE® in Healthy Volunteers
Brief Title: ADASUVE 2-dose Thorough QT/QTc Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: AMDC-204-407; 204-407 (Other: Alexza Pharmaceuticals, Inc)
Record Dates: First submitted 2013-05-08; First posted 2013-05-15 (Estimated); Results first posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2013-07

CONDITIONS: Healthy Volunteers
Keywords: ADASUVE; inhaled loxapine; thorough QT/QTc study
MeSH Terms: interventions — Loxapine; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, double-blind, double-dummy, 2-dose, 3-period, active- and placebo-controlled, crossover QT/QTc and pharmacokinetic (PK) study of ADASUVE in healthy volunteers. All dosing and treatment-day follow-up in the study was conducted in the clinical research unit (CRU)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Treatment sequence ABC (Other): Treatment: A = Inhaled loxapine (2 doses of 10 mg 2 hours apart) + oral placebo, B = Inhaled placebo + oral placebo, C = Oral moxifloxacin 400 mg + Inhaled placebo
  Interventions: Drug: ADASUVE 10 mg 2 doses 2 hours apart; Drug: Inhaled Placebo; Drug: Oral moxifloxacin 400 mg; Drug: Oral placebo
- Treatment sequence ACB (Other): Treatment: A = Inhaled loxapine (2 doses of 10 mg 2 hours apart) + oral placebo, B = Inhaled placebo + oral placebo, C = Oral moxifloxacin 400 mg + Inhaled placebo
  Interventions: Drug: ADASUVE 10 mg 2 doses 2 hours apart; Drug: Inhaled Placebo; Drug: Oral moxifloxacin 400 mg; Drug: Oral placebo
- Treatment sequence BCA (Other): Treatment: A = Inhaled loxapine (2 doses of 10 mg 2 hours apart) + oral placebo, B = Inhaled placebo + oral placebo, C = Oral moxifloxacin 400 mg + Inhaled placebo
  Interventions: Drug: ADASUVE 10 mg 2 doses 2 hours apart; Drug: Inhaled Placebo; Drug: Oral moxifloxacin 400 mg; Drug: Oral placebo
- Treatment sequence BAC (Other): Treatment: A = Inhaled loxapine (2 doses of 10 mg 2 hours apart) + oral placebo, B = Inhaled placebo + oral placebo, C = Oral moxifloxacin 400 mg + Inhaled placebo
  Interventions: Drug: ADASUVE 10 mg 2 doses 2 hours apart; Drug: Inhaled Placebo; Drug: Oral moxifloxacin 400 mg; Drug: Oral placebo
- Treatment sequence CAB (Other): Treatment: A = Inhaled loxapine (2 doses of 10 mg 2 hours apart) + oral placebo, B = Inhaled placebo + oral placebo, C = Oral moxifloxacin 400 mg + Inhaled placebo
  Interventions: Drug: ADASUVE 10 mg 2 doses 2 hours apart; Drug: Inhaled Placebo; Drug: Oral moxifloxacin 400 mg; Drug: Oral placebo
- Treatment sequence CBA (Other): Treatment: A = Inhaled loxapine (2 doses of 10 mg 2 hours apart) + oral placebo, B = Inhaled placebo + oral placebo, C = Oral moxifloxacin 400 mg + Inhaled placebo
  Interventions: Drug: ADASUVE 10 mg 2 doses 2 hours apart; Drug: Inhaled Placebo; Drug: Oral moxifloxacin 400 mg; Drug: Oral placebo

INTERVENTIONS:
Drug: ADASUVE 10 mg 2 doses 2 hours apart — Inhaled loxapine 10 mg 2 doses 2 hours apart
  Other Names: Staccato Loxapine
Drug: Inhaled Placebo — Staccato placebo via inhalation x 2 at 2 hours apart
Drug: Oral moxifloxacin 400 mg — Oral moxifloxacin 400 mg single dose
  Other Names: AVELOX
Drug: Oral placebo — Oral capsule identical in appearance to moxifloxacin

SUMMARY:
Assess the potential effects on the QT interval of 2 consecutive doses of ADASUVE administered 2 hours apart, in relation to placebo and an active control in healthy volunteers.

DETAILED DESCRIPTION:
It has been shown in a pre-marketing clinical study that clinically relevant QT prolongation does not appear to be associated with a single dose of ADASUVE. The potential risk of QTc prolongation following repeat dosing is unknown. Therefore the current study will assess the potential effects on the QT interval of 2 consecutive doses of ADASUVE administered 2 hours apart, in relation to placebo and an active control in healthy volunteers.

The study hypothesis H0: Placebo-subtracted max mean dQTc > 10 msec

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the ages of 18 to 65 years, inclusive.
* Body mass index (BMI) ≥18 and ≤32.
* Subjects who are willing and able to comply with the study schedule and requirements, and stay at the CRU for a 4-day period and 2 consecutive 3-day periods.
* Subjects who speak, read, and understand English and/or Dutch and are willing and able to provide written informed consent on an IEC approved form prior to the initiation of any study procedures.
* Subjects who are in good general health prior to study participation
* Female or male participants who agree to use a medically acceptable and effective birth control method

Exclusion Criteria:

* Subjects who regularly consume large amounts of xanthine-containing substances (≥ 5 cups of coffee/day).
* Subjects who have taken prescription or nonprescription medication within 5 days of Visit 2.
* Subjects who have had an acute illness within the last 5 days of Visit 2.
* Subjects who have smoked tobacco within the last 30 days or who have a positive cotinine test.
* Subjects who have a history of HIV, anti-HCV or HbsAg positivity.
* Subjects who have a history within the past 2 years of drug or alcohol dependence or abuse as defined by DSM-IV.
* Subjects who test positive for alcohol or have a positive urine drug screen.
* Subjects who have a history of allergy or intolerance to loxapine or amoxapine or history of bronchospasm following inhaled loxapine treatment.
* Subjects who have an ECG abnormality.
* Subjects who have hypotension, or hypertension.
* Subjects who have a history of unstable angina, syncope, coronary artery disease, myocardial infarction, congestive heart failure, transient ischemic attack, history of convulsions or other neurological disorder.
* Subjects who have a current history of asthma, chronic obstructive lung disease, or any other lung disease associated with bronchospasm.
* Subjects who use medications to treat airways disease, such as asthma or COPD.
* Subjects who have any acute respiratory signs/symptoms (e.g., wheezing).
* Female subjects who have a positive pregnancy test at screening or at admission to any of the treatment visits, or are breastfeeding.
* Subjects who have received an investigational drug within 60 days prior to the Screening Visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Nunes, MD, Principal Investigator — PRA Health Sciences
Locations (1):
- PRA International, Zuidlaren, Netherlands

IPD SHARING:
Plan to Share IPD: No
IPD submitted to regulatory authorities. Others may contact Alexza Pharmaceuticals, Inc. Please send your request to ClinicalTrialsInfo@alexza.com

REFERENCES:
- [Background] Cassella JV, Spyker DA, Yeung PP. A randomized, placebo-controlled repeat-dose thorough QT study of inhaled loxapine in healthy volunteers. Int J Clin Pharmacol Ther. 2015 Nov;53(11):963-71. doi: 10.5414/CP202457. PMID 26501204
- [Derived] Cassella JV, Spyker DA, Yeung PP. A randomized, placebo-controlled repeat-dose thorough QT study of inhaled loxapine in healthy volunteers. Int J Clin Pharmacol Ther. 2015 Oct 7. doi: 10.5414/CP202457. Online ahead of print. PMID 26445139

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Sequence ABC | Treatment Sequence ACB | Treatment Sequence BCA | Treatment Sequence BAC | Treatment Sequence CAB | Treatment Sequence CBA
Started | 10 | 10 | 10 | 10 | 10 | 10
Completed | 6 | 7 | 8 | 8 | 8 | 8
Not Completed | 4 | 3 | 2 | 2 | 2 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0 | 0 | 0
Not completed — CRI procedural error | 2 | 2 | 2 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population (N=60)
Groups:
- All Subjects Treated: All 6 treatment sequences = Safety Population
Arm/Group | All Subjects Treated
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (14.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 31
Region of Enrollment [Number; unit: participants]
  Netherlands | 60

OUTCOME MEASURES:

1. Primary Outcome: Maximum Effect of ADASUVE on Cardiac Repolarization (QTc Interval Duration) at the Maximum Clinical Dose Compared to Placebo
Description: Time-matched differences in QTcI values between the maximum of the mean difference from baseline of the QTcI interval after time-matched placebo subtraction for ADASUVE treatment at 12 post-inhalation times.
Time Frame: Predose, 2 min, 1, 1.5 hr, 2 hr 2 min, 2 hr 5 min, 2.5, 3, 5, 8, 12, and 24 hr
Population: QT population -- LSM and CI statistics were based on the individual (within subject) corrected differences between Adasuve and placebo exposures per ICH Guideline E14 for a thorough QT study.
Measure: Least Squares Mean (95% Confidence Interval); unit: msec
Groups:
- ADASUVE-Placebo Crossover Subjects: All subjects who completed both treatments A and B: Treatment: A = Inhaled loxapine (2 doses of 10 mg 2 hours apart) + oral placebo, B = Inhaled placebo + oral placebo.
  The analyses are based on a within (paired) comparison of the time matched drug - placebo QTc values.
Arm/Group | ADASUVE-Placebo Crossover Subjects
Number analyzed (Participants) | 44
msec | 4.04 [1.77 to 6.31]

2. Secondary Outcome: QTc Versus Loxapine Concentration
Description: QTc @ Cmax based on linear and nonlinear regression of QTcI versus time matched serum loxapine concentrations
Time Frame: Predose, 2 min, 1, 1.5 hr, 2 hr 2 min, 2 hr 5 min, 2.5, 3, 5, 8, 12, and 24 hr
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: msec
Groups:
- ADASUVE 10 mg x 2 Doses: ADASUVE QTcI, Differences from Placebo in Change from Pre-dose Baseline and One-sided 95% Upper Confidence Bound (msec)
  QTcI associated with mean Cmax
Arm/Group | ADASUVE 10 mg x 2 Doses
Number analyzed (Participants) | 44
msec | 2.6 [1.2 to 4.1]

3. Secondary Outcome: Subjects With QTcI > 450 ms
Description: Numbers of Subjects with QTcI > 450 ms at any time point
Time Frame: Predose, 2 min, 1, 1.5 hr, 2 hr 2 min, 2 hr 5 min, 2.5, 3, 5, 8, 12, and 24 hr
Population: QT population -- Comparisons were based on corrected differences between Adasuve and placebo (excluding moxifloxacin) exposure per ICH Guideline E14 for a thorough QT study.
Measure: Count of Participants; unit: Participants
Groups:
- Inhaled Placebo + Oral Placebo: Staccato Placebo 2 doses 2 hours apart + Oral Placebo
  Staccato Placebo 2 doses 2 hours apart: Inhaler with no drug in it to mimic the ADASUVE inhaler
  Placebo (for moxifloxacin): placebo capsule to mimic moxifloxacin 400 mg
- ADASUVE 10 mg x 2 Doses: ADASUVE 10 mg 2 doses 2 hours apart + Oral Placebo
  ADASUVE 10 mg 2 doses 2 hours apart: inhaled loxapine
  Placebo (for moxifloxacin): placebo capsule to mimic moxifloxacin 400 mg
Arm/Group | Inhaled Placebo + Oral Placebo | ADASUVE 10 mg x 2 Doses
Number analyzed (Participants) | 44 | 44
Participants | 2 | 2

4. Secondary Outcome: Subjects With QTcI > 480 ms
Description: Numbers of Subjects with QTcI > 480 ms (or 500 ms) at any time point
Time Frame: Predose, 2 min, 1, 1.5 hr, 2 hr 2 min, 2 hr 5 min, 2.5, 3, 5, 8, 12, and 24 hr
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Placebo + Oral Placebo | ADASUVE 10 mg x 2 Doses
Number analyzed (Participants) | 44 | 44
Participants | 0 | 0

5. Secondary Outcome: Subjects With QTcI Increase > 30 ms From Baseline
Description: Numbers of Subjects with QTcI Increase > 30 ms from Baseline at any time point
Time Frame: Predose, 2 min, 1, 1.5 hr, 2 hr 2 min, 2 hr 5 min, 2.5, 3, 5, 8, 12, and 24 hr
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Placebo + Oral Placebo | ADASUVE 10 mg x 2 Doses
Number analyzed (Participants) | 44 | 44
Participants | 0 | 1

6. Secondary Outcome: Subjects With QTcI Increase > 60 ms From Baseline
Description: Numbers of Subjects with QTcI Increase > 60 ms From Baseline at any time point
Time Frame: Predose, 2 min, 1, 1.5 hr, 2 hr 2 min, 2 hr 5 min, 2.5, 3, 5, 8, 12, and 24 hr
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Placebo + Oral Placebo | ADASUVE 10 mg x 2 Doses
Number analyzed (Participants) | 44 | 44
Participants | 0 | 0

7. Other Pre Specified Outcome: Maximum Effect of Moxifloxacin on Cardiac Repolarization (QTc Interval Duration) Compared to Placebo (Study Assay Sensitivity)
Description: A thorough QT/QTc study may be considered to have demonstrated assay sensitivity if 1 or more of the lower 95% CI values exceeds 5 msec
Time Frame: Predose, 2 min, 1, 1.5 hr, 2 hr 2 min, 2 hr 5 min, 2.5, 3, 5, 8, 12, and 24 hr
Population: QT population -- LSM and CI statistics were based on the individual (within subject) corrected differences between moxifloxacin and placebo exposures per ICH Guideline E14 for a thorough QT study.
Measure: Least Squares Mean (95% Confidence Interval); unit: msec
Groups:
- Moxifloxacin QT Crossover Subjects: All subjects who completed both Treatments B and C: B = Inhaled placebo + oral placebo, C = Oral moxifloxacin 400 mg + Inhaled placebo.
  Analyses are based on a within (paired) comparison of the time matched drug - placebo QTc values.
Arm/Group | Moxifloxacin QT Crossover Subjects
Number analyzed (Participants) | 44
msec | 10.47 [8.13 to 12.81]

ADVERSE EVENTS:
Time Frame: From first exposure to study treatment to 30 days after last exposure to study treatment
Description: Adverse events (AEs) were assessed pre-dose and at 12 prespecified time points
Groups:
- Oral Moxifloxacin: Staccato Placebo 2 doses 2 hours apart + Oral moxifloxacin 400 mg
  Oral moxifloxacin 400 mg
  Staccato Placebo 2 doses 2 hours apart: Inhaler with no drug in it to mimic the ADASUVE inhaler
Arm/Group | Inhaled Placebo + Oral Placebo | ADASUVE 10 mg x 2 Doses | Oral Moxifloxacin
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/52 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/52 | 0/49
Other Adverse Events (participants affected / at risk) | 15/49 | 38/52 | 9/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Placebo + Oral Placebo (N=49) | ADASUVE 10 mg x 2 Doses (N=52) | Oral Moxifloxacin (N=49)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0)
Dysgeusia (Gastrointestinal disorders) | 3 (3) | 8 (8) | 2 (2)
Fatigue (General disorders) | 2 (2) | 13 (13) | 2 (2)
Dizziness (Nervous system disorders) | 4 (4) | 12 (12) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 3 (3) | 2 (2)
Sedation (Nervous system disorders) | 4 (4) | 14 (14) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1) | 5 (5) | 1 (1)

LIMITATIONS AND CAVEATS:
The use of healthy subjects, which precludes observation of drug-induced QTc prolongation in a population with additional factors predisposing to TdP. Subjects with respiratory disease were excluded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less